CLINICAL TRIAL: NCT02514174
Title: A Single Arm Phase IV Study of Afatinib in Elderly Patients With Stage IV or Recurrent Non-Small Cell Lung Cancer Whose Tumors Have Epidermal Growth Factor Receptor (EGFR) Exon 19 Deletions or Exon 21(L858R) Substitution Mutations
Brief Title: Afatinib Treatment for Patients With EGFR Mutation Positive NSCLC Who Are Age 70 or Older
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1200.209
Record Dates: First submitted 2015-07-17; First posted 2015-08-03 (Estimated); Results first posted 2020-03-30 (Actual); Last update posted 2020-03-30 (Actual); Status verified 2020-03

CONDITIONS: Carcinoma, Non-Small-Cell Lung; ErbB Receptors
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Afatinib

ARMS (1):
- Afatinib (Experimental): afatinib starting at 30 mg daily dose
  Interventions: Drug: Afatinib

INTERVENTIONS:
Drug: Afatinib — afatinib starting at 30 mg daily dose

SUMMARY:
Continuous treatment until progression or occurence of intolerable Adverse Event (AE) or end of trial. The end of trial is one year after the last patient has entered the study.

ELIGIBILITY:
Inclusion criteria:

* Pathologically or cytologically confirmed NSCLC Stage IV Cancer (includes cytologically proven pleural effusion or pericardial effusion) or recurrent disease. Staging is based on American Joint Committee on Cancer (AJCC) Staging for NSCLC 7th edition (R12-4710)
* Evidence of common EGFR mutation (Del 19 and/or L858R)
* Age >= 70 years
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1 (R01-0787)
* Further inclusion criteria apply.

Exclusion criteria:

* Prior participation in an afatinib clinical study, even if not assigned to afatinib treatment
* Prior systemic therapy for metastatic or recurrent NSCLC.
* Concurrent investigational therapy or investigational therapy within 4 weeks of start of afatinib therapy
* Radiotherapy within 4 weeks prior to start of study treatment, except as follows:

  * Palliative radiation to target organs other than chest may be allowed up to 2 weeks prior to study treatment, or
  * Single dose palliative treatment for symptomatic metastasis outside above allowance to be discussed with sponsor prior to enrolling.
  * Major surgery within 4 weeks before starting study treatment or scheduled for surgery during the projected course of the study
  * Systemic chemotherapy, biological therapy, immunotherapy or investigational agents within 5 half-life of the drug or within four weeks prior to the start of afatinib treatment (if the half-life of the drug is unknown).
* Men, capable of fathering a child, who are unwilling to use adequate contraception prior to study entry, for the duration of study participation, and for at least 28 days after treatment has ended.
* Further exclusion criteria apply.

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 25 (Actual)
Dates: Start 2015-08-18 (Actual); Primary Completion 2019-03-28 (Actual); Study Completion 2019-04-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (10):
- United States (10):
  - Mayo Clinic-Arizona, Scottsdale, Arizona
  - Pacific Cancer Medical Center, Inc., Anaheim, California
  - City of Hope, Duarte, California
  - Compassionate Care Research Group, Inc. at Compassionate Cancer Care Medical Group, Inc., Fountain Valley, California
  - Los Angeles Hematology Oncology Medical Group, Los Angeles, California
  - University of Miami, Miami, Florida
  - Ingalls Memorial Hospital, Harvey, Illinois
  - Baystate Health D'Amour Center for Cancer Care, Springfield, Massachusetts
  - Montefiore Medical Center, The Bronx, New York
  - Lankenau Medical Center, Wynnewood, Pennsylvania

REFERENCES:
- See also: Related Info — https://trials.boehringer-ingelheim.com/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Open-label, non-randomized, Phase IV, single arm study
Pre-assignment Details: All subjects were screened for eligibility prior to participation in the trial. Subjects attended a specialist site which ensured that they (the subjects) strictly met all inclusion and none of the exclusion criteria. Subjects were not to be allocated to a treatment group if any of the entry criteria were violated.
Groups:
- Afatinib: Giotrif® / Gilotrif® (Afatinib) starting at 30 mg daily dose
  All participants received the same treatment (afatinib) with starting dose of 30 milligram (mg) per day with one possible dose reduction to 20 mg per day.
  Mode of administration: Orally one film-coated tablet, once daily
Period: Overall Study
Arm/Group | Afatinib
Started ((Participants who were dispensed afatinib and were documented to have taken at least one dose.)) | 25
Completed | 0
Not Completed | 25
Not completed — Patient refused to continue medication | 1
Not completed — Adverse Event | 2
Not completed — Study closed by sponsor | 9
Not completed — Progressive disease | 11
Not completed — Treatment change | 1
Not completed — Treated off study with Afatinib. | 1

BASELINE CHARACTERISTICS:
Population: All participants who received at least one dose of afatinib were included in the treated set. The analyses of safety and efficacy were performed on the treated set.
Arm/Group | Afatinib
Number analyzed (Participants) | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 79.2 (5.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 22
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 8
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 14
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Reporting an Adverse Event (AE) Leading to Dose Reduction of Afatinib
Description: On-treatment period = First administration of afatinib until progression or intolerable adverse events or other reasons necessitating withdrawal (participant's withdrawal of consent for study treatment, participant diagnosed with interstitial lung disease, participant no longer able to receive study treatments, participant had a significant deviation from the protocol or eligibility criteria).
Time Frame: On-treatment period + 28 days (residual effect period), up to 1057 + 28 days
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: Percentage
Arm/Group | Afatinib
Number analyzed (Participants) | 25
Percentage | 32.0 [14.9 to 53.5]

2. Secondary Outcome: Percentage of Participants With Adverse Event = Diarrhoea of Common Terminology Criteria for Adverse Events (CTCAE) Grade 3 or Higher
Description: Percentage of participants with adverse event being diarrhoea of CTCAE grade 3 or higher.
  On-treatment period = First administration of afatinib until progression or intolerable adverse events or other reasons necessitating withdrawal (participant's withdrawal of consent for study treatment, participant diagnosed with interstitial lung disease, participant no longer able to receive study treatments, participant had a significant deviation from the protocol or eligibility criteria).
Time Frame: On-treatment period + 28 days (residual effect period), up to 1057 + 28 days
Population: as for baseline characteristics
Measure: Number; unit: Percentage of participants
Arm/Group | Afatinib
Number analyzed (Participants) | 25
Percentage of participants | 8.0

3. Secondary Outcome: Percentage of Participants With Adverse Event = Rash/Acne (Grouped Term) of CTCAE Grade 3 or Higher
Description: Percentage of participants with adverse event = rash/acne (grouped term) of CTCAE grade 3 or higher.
  MedDRA preferred terms that described AEs of similar nature were grouped together as "grouped term" to ensure that important events would not be underestimated.
  On-treatment period = First administration of afatinib until progression or intolerable adverse events or other reasons necessitating withdrawal (participant's withdrawal of consent for study treatment, participant diagnosed with interstitial lung disease, participant no longer able to receive study treatments, participant had a significant deviation from the protocol or eligibility criteria).
Time Frame: On-treatment period + 28 days (residual effect period), up to 1057 + 28 days
Population: as for baseline characteristics
Measure: Number; unit: Percentage of participants
Arm/Group | Afatinib
Number analyzed (Participants) | 25
Percentage of participants | 0.0

4. Secondary Outcome: Percentage of Participants With Adverse Event = Stomatitis (Grouped Term) of CTCAE Grade 3 or Higher
Description: Percentage of participants with adverse event = stomatitis (grouped term) of CTCAE grade 3 or higher.
  MedDRA preferred terms that described AEs of similar nature were grouped together as "grouped term" to ensure that important events would not be underestimated.
  On-treatment period = First administration of afatinib until progression or intolerable adverse events or other reasons necessitating withdrawal (participant's withdrawal of consent for study treatment, participant diagnosed with interstitial lung disease, participant no longer able to receive study treatments, participant had a significant deviation from the protocol or eligibility criteria).
Time Frame: On-treatment period + 28 days (residual effect period), up to 1057 + 28 days
Population: as for baseline characteristics
Measure: Number; unit: Percentage of participants
Arm/Group | Afatinib
Number analyzed (Participants) | 25
Percentage of participants | 4.0

5. Secondary Outcome: Percentage of Participants With Adverse Event = Paronychia (Grouped Term) of CTCAE Grade 3 or Higher
Description: Percentage of participants with adverse event = paronychia (grouped term) of CTCAE grade 3 or higher.
  MedDRA preferred terms that described AEs of similar nature were grouped together as "grouped term" to ensure that important events would not be underestimated.
  On-treatment period = First administration of afatinib until progression or intolerable adverse events or other reasons necessitating withdrawal (participant's withdrawal of consent for study treatment, participant diagnosed with interstitial lung disease, participant no longer able to receive study treatments, participant had a significant deviation from the protocol or eligibility criteria).
Time Frame: On-treatment period + 28 days (residual effect period), up to 1057 + 28 days
Population: as for baseline characteristics
Measure: Number; unit: Percentage of participants
Arm/Group | Afatinib
Number analyzed (Participants) | 25
Percentage of participants | 8.0

6. Secondary Outcome: Time to First Dose Reduction of Afatinib Caused by Adverse Events
Description: Time to first dose reduction of afatinib caused by adverse events is defined as time from the date of the first administration of afatinib to the date of first dose reduction of afatinib caused by adverse events. Participants without AEs leading to dose reduction were censored at date of last intake of afatinib.
  On-treatment period = First administration of afatinib until progression or intolerable adverse events or other reasons necessitating withdrawal (participant's withdrawal of consent from study treatment, participant diagnosed with interstitial lung disease, participant no longer able to receive study treatments, participant had a significant deviation from the protocol or eligibility criteria).
  The cumulative probability of no dose reduction at the respective time point is given by the Kaplan-Meier estimate at the respective time point based on time to first dose reduction of afatinib caused by adverse events.
Time Frame: On-treatment period, up to 1057 days
Population: All participants who received at least one dose of afatinib were included in the treated set. The analyses of safety and efficacy were performed on the treated set.
  The 'Number Analyzed' is the 'Number at risk' at the respective time point, that is the number of participants being treated with afatinib 30 mg at the respective time point.
Measure: Number (95% Confidence Interval); unit: Probability
Arm/Group | Afatinib
Number analyzed (Participants) | 25
Probability
  0 months (= First administration of afatinib) | 1.0 [1.0 to 1.0]
  3 months: number analyzed (Participants) | 18
  3 months | 0.7889 [0.5642 to 0.9064]
  6 months: number analyzed (Participants) | 18
  6 months | 0.7450 [0.5176 to 0.8768]
  9 months: number analyzed (Participants) | 13
  9 months | 0.6519 [0.4214 to 0.8091]
  12 months: number analyzed (Participants) | 12
  12 months | 0.6519 [0.4214 to 0.8091]
  15 months: number analyzed (Participants) | 9
  15 months | 0.6519 [0.4214 to 0.8091]
  18 months: number analyzed (Participants) | 6
  18 months | 0.6519 [0.4214 to 0.8091]
  21 months: number analyzed (Participants) | 5
  21 months | 0.6519 [0.4214 to 0.8091]
  24 months: number analyzed (Participants) | 5
  24 months | 0.6519 [0.4214 to 0.8091]
  27 months: number analyzed (Participants) | 2
  27 months | 0.6519 [0.4214 to 0.8091]
  30 months: number analyzed (Participants) | 1
  30 months | 0.6519 [0.4214 to 0.8091]
  33 months: number analyzed (Participants) | 1
  33 months | 0.6519 [0.4214 to 0.8091]

ADVERSE EVENTS:
Time Frame: On-treatment period+28 days, up to 1057+28 days. On-treatment period=First administration of afatinib until progression or intolerable AEs or other reasons necessitating withdrawal (participant withdrew consent or was diagnosed with interstitial lung disease or was no longer able to receive study treatments or had a significant deviation from the protocol or eligibility criteria). Time Frame for All-Cause Mortality is On-treatment period + Follow-Up, up to 1096 days.
Description: Adverse events (AEs) were reported for the treated set which comprises all participants who received at least one dose of afatinib.
  From 28 days after last trial drug intake new AEs were only reported if they were considered related to trial drug.
Groups:
- Afatinib 30 mg: Giotrif® / Gilotrif® (Afatinib) starting at 30 mg daily dose
  All participants received the same treatment (afatinib) with starting dose of 30 milligram (mg) per day with one possible dose reduction to 20 mg per day.
  Mode of administration: Orally one film-coated tablet, once daily
Arm/Group | Afatinib 30 mg
All-Cause Mortality (participants affected / at risk) | 7/25
Serious Adverse Events (participants affected / at risk) | 10/25
Other Adverse Events (participants affected / at risk) | 25/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Afatinib 30 mg (N=25)
Diarrhoea (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Rectal haemorrhage (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 2
Pneumonia (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Fall (Injury, poisoning and procedural complications) | 1
Fracture displacement (Injury, poisoning and procedural complications) | 1
Humerus fracture (Injury, poisoning and procedural complications) | 1
Joint dislocation (Injury, poisoning and procedural complications) | 1
Dehydration (Metabolism and nutrition disorders) | 2
Hyponatraemia (Metabolism and nutrition disorders) | 1
Hypovolaemia (Metabolism and nutrition disorders) | 1
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Seizure (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 2
Acute kidney injury (Renal and urinary disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Afatinib 30 mg (N=25)
Anaemia (Blood and lymphatic system disorders) | 2
Dry eye (Eye disorders) | 7
Vision blurred (Eye disorders) | 2
Abdominal pain (Gastrointestinal disorders) | 2
Abdominal pain upper (Gastrointestinal disorders) | 3
Constipation (Gastrointestinal disorders) | 6
Diarrhoea (Gastrointestinal disorders) | 22
Dry mouth (Gastrointestinal disorders) | 8
Dyspepsia (Gastrointestinal disorders) | 3
Haemorrhoids (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 9
Oral pain (Gastrointestinal disorders) | 2
Proctalgia (Gastrointestinal disorders) | 2
Rectal haemorrhage (Gastrointestinal disorders) | 2
Stomatitis (Gastrointestinal disorders) | 9
Vomiting (Gastrointestinal disorders) | 6
Chills (General disorders) | 2
Fatigue (General disorders) | 12
Gait disturbance (General disorders) | 2
Non-cardiac chest pain (General disorders) | 3
Oedema (General disorders) | 2
Oedema peripheral (General disorders) | 3
Pain (General disorders) | 4
Pyrexia (General disorders) | 2
Bronchitis (Infections and infestations) | 2
Conjunctivitis (Infections and infestations) | 2
Fungal skin infection (Infections and infestations) | 2
Nail infection (Infections and infestations) | 2
Paronychia (Infections and infestations) | 6
Pneumonia (Infections and infestations) | 3
Sinusitis (Infections and infestations) | 3
Upper respiratory tract infection (Infections and infestations) | 8
Urinary tract infection (Infections and infestations) | 4
Contusion (Injury, poisoning and procedural complications) | 2
Skin abrasion (Injury, poisoning and procedural complications) | 2
Weight decreased (Investigations) | 3
Decreased appetite (Metabolism and nutrition disorders) | 8
Dehydration (Metabolism and nutrition disorders) | 3
Hypokalaemia (Metabolism and nutrition disorders) | 4
Hypomagnesaemia (Metabolism and nutrition disorders) | 3
Hyponatraemia (Metabolism and nutrition disorders) | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 4
Back pain (Musculoskeletal and connective tissue disorders) | 7
Flank pain (Musculoskeletal and connective tissue disorders) | 2
Joint swelling (Musculoskeletal and connective tissue disorders) | 3
Muscle spasms (Musculoskeletal and connective tissue disorders) | 5
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3
Dizziness (Nervous system disorders) | 4
Headache (Nervous system disorders) | 4
Hypoaesthesia (Nervous system disorders) | 2
Neuropathy peripheral (Nervous system disorders) | 3
Paraesthesia (Nervous system disorders) | 2
Anxiety (Psychiatric disorders) | 2
Insomnia (Psychiatric disorders) | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 7
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 8
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 2
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 5
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3
Productive cough (Respiratory, thoracic and mediastinal disorders) | 3
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 2
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 2
Alopecia (Skin and subcutaneous tissue disorders) | 5
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 4
Dry skin (Skin and subcutaneous tissue disorders) | 13
Erythema (Skin and subcutaneous tissue disorders) | 2
Hair texture abnormal (Skin and subcutaneous tissue disorders) | 2
Nail discolouration (Skin and subcutaneous tissue disorders) | 2
Onychoclasis (Skin and subcutaneous tissue disorders) | 7
Pruritus (Skin and subcutaneous tissue disorders) | 4
Rash (Skin and subcutaneous tissue disorders) | 16
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 5
Scab (Skin and subcutaneous tissue disorders) | 2
Skin atrophy (Skin and subcutaneous tissue disorders) | 2
Skin discolouration (Skin and subcutaneous tissue disorders) | 2
Skin exfoliation (Skin and subcutaneous tissue disorders) | 3
Skin fissures (Skin and subcutaneous tissue disorders) | 3

LIMITATIONS AND CAVEATS:
Limitation: Protocol was amended on 15-February-2018 to reduce total sample size from n=50 participants to n=25 participants due to slow enrollment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The rights of the investigator and of the sponsor with regard to publication of the results of this trial were described in a separate agreement between the investigator or the trial site and the sponsor. As a general rule, no trial results were to be published prior to finalization of the clinical trial report.

DOCUMENTS (2):
  • Study Protocol (2018-02-15): https://cdn.clinicaltrials.gov/large-docs/74/NCT02514174/Prot_000.pdf
  • Statistical Analysis Plan (2019-03-25): https://cdn.clinicaltrials.gov/large-docs/74/NCT02514174/SAP_001.pdf